CLINICAL TRIAL: NCT00812240
Title: A Prospective, Multicenter, Randomized, Open-label, Active-controlled, 2-parallel Group, Phase III Study to Compare Efficacy and Safety of Masitinib at 7.5 mg/kg/Day to Imatinib at 400 or 600 mg in Treatment of Patients With Gastro-intestinal Stromal Tumor in First Line Medical Treatment
Brief Title: Masitinib in First Line Treatment of Gastro-Intestinal Stromal Tumor (GIST)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision based on portfolio prioritization
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB04030
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2023-02-01 (Actual); Status verified 2019-12

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastro-Intestinal Stromal Tumor; GIST; metastatic; non resectable locally advanced
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasm Metastasis | interventions — masitinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Masitinib (7.5) (Experimental): Participants receive masitinib (7.5 mg/kg/day), given orally twice daily.
  Interventions: Drug: Masitinib
- Masitinib (6.0) (Experimental): Participants receive masitinib (6.0 mg/kg/day), given orally twice daily
  Interventions: Drug: Masitinib
- Active Comparator (7.5) (Active Comparator): Participants receive imatinib at 400 or 600 mg per day
  Interventions: Drug: Imatinib
- Active Comparator (6.0) (Active Comparator): Participants receive imatinib at 400 or 600 mg per day
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Masitinib
  Other Names: AB1010
  Arms: Masitinib (6.0); Masitinib (7.5)
Drug: Imatinib — imatinib 400 mg or 600 mg per day, per os
  Other Names: Gleevec
  Arms: Active Comparator (6.0); Active Comparator (7.5)

SUMMARY:
Masitinib in First Line Treatment of Gastro-Intestinal Stromal Tumor (GIST)

DETAILED DESCRIPTION:
Masitinib is a selective tyrosine kinase inhibitor with potent activity against wild-type c-Kit, the juxta membrane domain of c-Kit, and PDGFR. In addition to its direct inhibitory action against these kinase targets, masitinib is also thought to promote survival via modulation of immunostimulation-mediated anticancer effects and modulation of the tumor microenvironment. The objective of this prospective, multicenter, randomized, open-label, active-controlled study is to compare the efficacy and safety of masitinib with respect to imatinib in the first line treatment of gastro-intestinal stromal tumor (GIST). Treatment will be given until disease progression, limiting toxicity or patient consent withdrawal.

ELIGIBILITY:
Main inclusion criteria include:

* Histologically proven, metastatic or locally advanced non resectable, or recurrent post-surgery GIST
* Naïve patient or patient previously treated with imatinib as neoadjuvant/adjuvant who relapsed after imatinib discontinuation
* c-Kit (CD117) positive tumours detected by immuno-histochemically or PDGFR positive if c-Kit negative

Main exclusion criteria include:

* Patient previously treated by tyrosine kinase inhibitors except imatinib in case of inclusion criteria
* Patient treated for a cancer other than GIST within 5 years before enrolment, with the exception of basal cell carcinoma or cervical cancer in situ
* Patient with active central nervous system (CNS) metastasis or with history of CNS metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From day of randomization to disease progression or death, assessed for a maximum of 96 months]
  Progression Free Survival is defined as the time from randomization to first documentation of objective tumor progression (date of tumor assessment documenting progressive disease assessed by CT Scan according to RECIST 1.1 and based on central review) or to death due to any cause (whichever comes first).

SECONDARY OUTCOMES:
Overall Survival (OS) | From day of randomization to death, assessed for a maximum of 96 months
  Overall survival is defined as time in months from the randomization date to the date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Adenis, MD, Principal Investigator — Centre Oscar Lambret, Lille, France
Locations (41):
- United States (7):
  - MD Anderson Cancer Center, Orlando, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Henry Ford Health System, Detroit, Michigan
  - Beth Israel Medical Center, New York, New York
  - Ohio State University, Columbus, Ohio
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- France (29):
  - Centre Hospitalier d'Abbeville, Abbeville
  - Institut Sainte Catherine, Avignon
  - Hôpital Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Hôpital Morvan, Brest
  - Hôpitalo Henri Mondor, Créteil
  - Centre Georges François Leclerc, Dijon
  - Hopital Bocage, Dijon
  - Centre Hospitalier Victor Jousselin, Dreux
  - Clinique Pasteur, Évreux
  - Centre Hospitalier de Gap, Gap
  - CHD de Vendée, La Roche-sur-Yon
  - Centre Hsopitalier de La Rochelle, La Rochelle
  - Centre Hospitalier Robert Boulin, Libourne
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmette, Marseille
  - Centre Val d'Aurèle, Montpellier
  - Centre René Gauducheau, Nantes
  - Hôpital de la Source, Orléans
  - Groupe Hospitalier Diaconesse Croix Saint Simon, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Bichat Claude Bernard, Paris
  - Hôpital Tenon, Paris
  - Hôpital Robert Debré, Reims
  - Hôpital Charles Nicolle, Rouen
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - Centre René Huguenin, Saint-Cloud
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
- Lebanon (5):
  - Hotel Dieu de France, Beirut
  - Hôpital Saint-Georges, Beirut
  - Makassed General Hospital Tarik Jadide, Beirut
  - Rafik Hariri University Hospital, Beirut
  - Hôpital Saint-Joseph, Jdeïdé